CLINICAL TRIAL: NCT04510103
Title: A Bilateral, Controlled Clinical Trial to Evaluate 2 Different Moisturizer Chassis Formulas for the Relief of Dry Skin
Brief Title: A Controlled Clinical Study of 2 Different Moisturizers for the Relief of Dry Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PS-150914160029-SACT
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Skin; Skin Care; Skin Cream
Keywords: Skin; Stratum Corneum; Skin Care; Skin Cream; Dryness; Moisturization; Hydration

STUDY DESIGN:
Intervention Model Description: Subjects were assigned to one of two procedural groups (Regression or Non-Regression) based on Visit 1 scheduling. Subjects were provided with a commercial cleanser to use during a 3-day period with no moisturizers and no hair removal allowed on their lower legs, and to continue using throughout the study. At Visit 2, all subjects received the two test moisturizers to use split-leg (right vs. left lower leg randomized) to use for 6 weeks. Subjects returned for evaluations at Week 2 (Visit 3), Week 4 (Visit 4), and Week 6 (Visit 5). At Week 6, subjects in the Regression group entered a 2-week regression period (no moisturizer usage) and returned for evaluations at Regression Days 1, 4, 7, 10, and 14. Meanwhile, at Week 6, subjects in the Non-Regression group (exploratory) continued using the moisturizers; they returned for evaluations at Week 6 + Days 1, 2, 3, and 4.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The test moisturizers were assigned a product code; each moisturizer was assigned to a subject's right or left lower leg per a randomization schedule. Subjects were blinded to the product identities, and evaluators were blinded to which product was used on each leg. Procedural group was unblinded and based on scheduling at Visit 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regression Group (Other): The Regression Group received the two test moisturizers to use split-leg (right vs. left lower leg randomized) for 6 weeks and then entered a 2-week regression period (no moisturizer usage).
  Interventions: Drug: Moisturizer A, F#9155-005; Other: Moisturizer B, F#E1387-004; Procedure: Regression
- Non-Regression Group (Other): The Non-Regression Group received the two test moisturizers to use split-leg (right vs. left lower leg randomized) for 6 weeks and then underwent a physical insult (tape stripping) on the lower legs and continued using the moisturizer for 4 additional days.
  Interventions: Drug: Moisturizer A, F#9155-005; Other: Moisturizer B, F#E1387-004; Procedure: Non-Regression

INTERVENTIONS:
Drug: Moisturizer A, F#9155-005 — OTC Monograph Drug. Used twice daily on left or right lower leg per randomization schedule.
Other: Moisturizer B, F#E1387-004 — Cosmetic Moisturizer. Used twice daily on left or right lower leg per randomization schedule.
Procedure: Regression — 2 week regression period after 6 weeks of moisturizer use.
  Arms: Regression Group
Procedure: Non-Regression — Physical insult (tape stripping) on the lower leg after 6 weeks of moisturizer use.
  Arms: Non-Regression Group

SUMMARY:
Dry skin is characterized by a lack of moisture in the outer layer of the skin and can occur as a result of numerous factors including cold weather, low humidity, age, etc. In this study, the moisturizing benefits of two formulas were evaluated for barrier function improvement/impact when used by women with moderately to severely dry skin on their lower legs.

ELIGIBILITY:
Inclusion Criteria:

* moderately to severely dry skin on both leg legs, as determined by the investigator.
* Fitzpatrick skin types I-IV
* generally in good health
* routinely uses moisturizers on the legs at least 1-3 times per week.
* if of reproductive potential: using a medically acceptable form of birth control for at least 3 months before the study and willing to continue it for at least 1 month after study completion.
* able to read, write, speak, and understand English.
* willing and able to complete all study instructions.
* has completed the informed consent document including a HIPAA disclosure and photograph release.

Exclusion Criteria:

* known allergies/sensitivities to adhesive tapes or study product ingredients.
* known skin conditions, uncontrolled medical conditions, or any other condition that could interfere with evaluations/data interpretation or increase risk to the subject.
* any active bacterial/fungal/viral skin infections or susceptibility to such infections.
* females who are pregnant, breastfeeding, or planning to become pregnant in near future.
* compromised/broken skin, tattoos, scarring, excessive hair growth, very uneven skin tone, or other conditions that would interfere with evaluations or increase risk to the subject.
* current participation in another study.
* participation in another study in past 4 weeks.
* employees or relatives of the investigator or study site.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline to Week 6 in Clinical Grading of Skin Dryness | Baseline to Week 6
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.

SECONDARY OUTCOMES:
Mean Change from Baseline to Week 2 in Clinical Grading of Skin Dryness | Baseline to Week 2
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Baseline to Week 4 in Clinical Grading of Skin Dryness | Baseline to Week 4
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Regression Baseline to Regression Day 1 in Clinical Grading of Skin Dryness | Regression Baseline to Regression Day 1
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Regression Baseline to Regression Day 4 in Clinical Grading of Skin Dryness | Regression Baseline to Regression Day 4
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Regression Baseline to Regression Day 7 in Clinical Grading of Skin Dryness | Regression Baseline to Regression Day 7
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Regression Baseline to Regression Day 10 in Clinical Grading of Skin Dryness | Regression Baseline to Regression Day 10
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Regression Baseline to Regression Day 14 in Clinical Grading of Skin Dryness | Regression Baseline to Regression Day 14
  The investigator assessed each of the subject's lower legs for skin dryness on a scale of 0 (no dryness) to 4 (severe scaling/fissuring). Half-points allowed.
Mean Change from Baseline to Week 2 in Clinical Grading of Skin Cracking | Baseline to Week 2
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Baseline to Week 4 in Clinical Grading of Skin Cracking | Baseline to Week 4
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Baseline to Week 6 in Clinical Grading of Skin Cracking | Baseline to Week 6
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Regression Baseline to Regression Day 1 in Clinical Grading of Skin Cracking | Regression Baseline to Regression Day 1
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Regression Baseline to Regression Day 4 in Clinical Grading of Skin Cracking | Regression Baseline to Regression Day 4
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Regression Baseline to Regression Day 7 in Clinical Grading of Skin Cracking | Regression Baseline to Regression Day 7
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Regression Baseline to Regression Day 10 in Clinical Grading of Skin Cracking | Regression Baseline to Regression Day 10
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Regression Baseline to Regression Day 14 in Clinical Grading of Skin Cracking | Regression Baseline to Regression Day 14
  The investigator assessed each of the subject's lower legs for skin cracking on a scale of 0 (none) to 8 (obvious cracking). Whole points only.
Mean Change from Baseline to Week 2 in Clinical Grading of Skin Scaling | Baseline to Week 2
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Baseline to Week 4 in Clinical Grading of Skin Scaling | Baseline to Week 4
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Baseline to Week 6 in Clinical Grading of Skin Scaling | Baseline to Week 6
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Regression Baseline to Regression Day 1 in Clinical Grading of Skin Scaling | Regression Baseline to Regression Day 1
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Regression Baseline to Regression Day 4 in Clinical Grading of Skin Scaling | Regression Baseline to Regression Day 4
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Regression Baseline to Regression Day 7 in Clinical Grading of Skin Scaling | Regression Baseline to Regression Day 7
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Regression Baseline to Regression Day 10 in Clinical Grading of Skin Scaling | Regression Baseline to Regression Day 10
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Regression Baseline to Regression Day 14 in Clinical Grading of Skin Scaling | Regression Baseline to Regression Day 14
  The investigator assessed each of the subject's lower legs for skin scaling on a scale of 0 (none) to 8 (large scales). Whole points only.
Mean Change from Baseline to Week 2 in Clinical Grading of Tactile Roughness | Baseline to Week 2
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Baseline to Week 4 in Clinical Grading of Tactile Roughness | Baseline to Week 4
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Baseline to Week 6 in Clinical Grading of Tactile Roughness | Baseline to Week 6
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Regression Baseline to Regression Day 1 in Clinical Grading of Tactile Roughness | Regression Baseline to Regression Day 1
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Regression Baseline to Regression Day 4 in Clinical Grading of Tactile Roughness | Regression Baseline to Regression Day 4
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Regression Baseline to Regression Day 7 in Clinical Grading of Tactile Roughness | Regression Baseline to Regression Day 7
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Regression Baseline to Regression Day 10 in Clinical Grading of Tactile Roughness | Regression Baseline to Regression Day 10
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Regression Baseline to Regression Day 14 in Clinical Grading of Tactile Roughness | Regression Baseline to Regression Day 14
  The investigator assessed each of the subject's lower legs for tactile roughness on a scale of 0 (none) to 3 (severe) scale. Half-points allowed.
Mean Change from Baseline to Week 2 in Clinical Tolerance Grading | Baseline to Week 2
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Baseline to Week 4 in Clinical Tolerance Grading | Baseline to Week 4
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Baseline to Week 6 in Clinical Tolerance Grading | Baseline to Week 6
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Regression Baseline to Regression Day 1 in Clinical Tolerance Grading | Regression Baseline to Regression Day 1
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Regression Baseline to Regression Day 4 in Clinical Tolerance Grading | Regression Baseline to Regression Day 4
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Regression Baseline to Regression Day 7 in Clinical Tolerance Grading | Regression Baseline to Regression Day 7
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Regression Baseline to Regression Day 10 in Clinical Tolerance Grading | Regression Baseline to Regression Day 10
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Regression Baseline to Regression Day 14 in Clinical Tolerance Grading | Regression Baseline to Regression Day 14
  The investigator assessed each of the subject's lower legs for the following tolerance parameters on a scale of 0 (none) to 3 (severe):
  * erythema
  * edema
  * burning/stinging (via subject interview)
  * itching (via subject interview)
  * tightness (via subject interview) Half-points allowed.
Mean Change from Baseline to Week 4 in TEWL | Baseline to Week 4
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Baseline to Week 6 in TEWL | Baseline to Week 6
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Regression Baseline to Regression Day 1 in TEWL | Regression Baseline to Regression Day 1
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Regression Baseline to Regression Day 4 in TEWL | Regression Baseline to Regression Day 4
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Regression Baseline to Regression Day 7 in TEWL | Regression Baseline to Regression Day 7
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Regression Baseline to Regression Day 10 in TEWL | Regression Baseline to Regression Day 10
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Regression Baseline to Regression Day 14 in TEWL | Regression Baseline to Regression Day 14
  Transepidermal water loss (TEWL), a measure of the passive transfer of water through the outer layer of the skin in g/m2/h, was measured with an open-chambered evaporimeter. Three measurements were taken per leg.
Mean Change from Baseline to Week 4 in Skin Hydration | Baseline to Week 4
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Baseline to Week 6 in Skin Hydration | Baseline to Week 6
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Regression Baseline to Regression Day 1 in Skin Hydration | Regression Baseline to Regression Day 1
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Regression Baseline to Regression Day 4 in Skin Hydration | Regression Baseline to Regression Day 4
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Regression Baseline to Regression Day 7 in Skin Hydration | Regression Baseline to Regression Day 7
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Regression Baseline to Regression Day 10 in Skin Hydration | Regression Baseline to Regression Day 10
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Regression Baseline to Regression Day 14 in Skin Hydration | Regression Baseline to Regression Day 14
  Skin hydration of the lower legs was measured with two different instruments: 1) a Corneometer, which measures hydration in arbitrary units from 0 to 120, with higher values indicating more hydrated skin, and 2) Skicon, which measures hydration in microSiemens (uS) from 0 to 2000, with higher values indicating more hydrated skin. Five measurements were taken with each instrument.
Mean Change from Baseline to Week 4 in Skin Flaking using D-Squames | Baseline to Week 4
  D-Squame tapes were used to collect skin surface cells. The first tape was placed on a D-Squame storage card. Image analysis was used to calculate the degree of skin flaking.
Mean Change from Baseline to Week 6 in Skin Flaking using D-Squames | Baseline to Week 6
  D-Squame tapes were used to collect skin surface cells. The first tape was placed on a D-Squame storage card. Image analysis was used to calculate the degree of skin flaking.
Mean Change from Baseline to Week 4 in NMFs using D-Squames | Baseline to Week 4
  D-Squame tapes were used to collect skin surface cells. The second tape was stored in a scintillation vial and shipped to a designated lab for analysis of natural moisturizing factors (NMFs), components of the skin that help it maintain adequate hydration.
Mean Change from Baseline to Week 6 in NMFs using D-Squames | Baseline to Week 6
  D-Squame tapes were used to collect skin surface cells. The second tape was stored in a scintillation vial and shipped to a designated lab for analysis of natural moisturizing factors (NMFs), components of the skin that help it maintain adequate hydration.
Mean Change from Baseline to Week 4 in Epidermal Lipids | Baseline to Week 4
  Special adhesive tapes were used to collect and analyze epidermal lipid samples from the skin surface.
Mean Change from Baseline to Week 6 in Epidermal Lipids | Baseline to Week 6
  Special adhesive tapes were used to collect and analyze epidermal lipid samples from the skin surface.

CONTACTS AND LOCATIONS:
Overall Officials: Neena Tierney, Study Director — Johnson & Johnson Consumer Inc. (J&JCI); Kun "Mark" Qian, M.D., Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (1):
- Thomas J. Stephens & Associates, Inc., Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu